CLINICAL TRIAL: NCT04274699
Title: Clinical Evaluation of the Hemosonics Quantra® Coagulation Monitor in Liver and Multivisceral Transplantation
Status: Withdrawn | Type: Observational
Why Stopped: Funding withdrawn by commercial partner before recruitment phase (change of company ownership).
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: HemoSonics LLC (Industry)
Responsible Party: Principal Investigator, John Klinck, Consultant Anaesthetist, Principal Investigator, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A095196 IRAS_ID_256865
Record Dates: First submitted 2020-02-15; First posted 2020-02-18 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2020-02

CONDITIONS: Coagulopathy; Liver Transplantation
Keywords: Liver Transplantation; Thromboelastography; Coagulopathy
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Citrated blood for thrombin generation assay
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Hemosonics Quantra coagulation monitor — There is no categorisation or allocation of any subject to any intervention vs non-intervention group. Blood sampling and the addition of a Quantra coagulation test is the only 'intervention', and the sampling protocol is identical for all subjects. Post-testing treatment of all subjects is as per established routine and Quantra results will not be used by clinical team.

SUMMARY:
Severe coagulopathy and operative bleeding are common in liver and multivisceral transplant recipients. This is related to reduced synthesis and function of clotting proteins in end-stage liver disease, thrombocytopaenia, thrombocytopathy, accelerated fibrinolysis, portal hypertension, inflammatory adhesions and intraoperative hemodilution. A pro-coagulant state is also a common finding in both groups, sometimes associated with fatal thromboembolism, and the balance between anti- and pro-coagulant effects is easily disrupted by intraoperative events. Use of point-of-care intraoperative viscoelastic testing, capable of discriminating between various potential causes of coagulopathy and of identifying some hypercoagulable states, is now routine in this setting. This has been shown to guide treatment faster and more reliably than standard laboratory screening tests.

However, traditional viscoelastic tests based on a pin-and-cup arrangement are sensitive to technical error, movement and physical clot disruption, and the validity of measurements is highly dependent on operator training. A newer method (TEG® 6S) based on light reflection from a blood meniscus reduces scope for operator error but remains sensitive to movement. Measurement of ultrasonic resonance (or 'sonic estimation of elasticity via resonance [SEER] sonorheometry') using the Quantra® analyzer surgery appears to minimize these problems in studies performed in healthy volunteers, in spinal surgery and in both elective and urgent cardiac procedures. Pilot testing in the latter group suggests it may also differentiate qualitatively between fibrinogen and platelet deficiency, but the range of intrinsic coagulation disturbances in this context is limited. This study proposes to assess the validity of the Quantra® analyzer in a population with more extreme coagulopathy, including severe fibrinolysis, and recognized thrombophilic states.

DETAILED DESCRIPTION:
Blood clotting during surgery is a complex process affected by many factors, including low levels of clotting factors and/or platelets resulting from liver disease, varying levels of factors that promote clotting, medicines that inhibit clotting, dilution of clotting factors by fluids given during surgery, body temperature, haemoglobin levels, inflammation, and tissue factors that speed up the breakdown of newly formed clots. The treatment of excessive surgical bleeding and abnormal clotting (thrombosis) depends on distinguishing between these factors to target the probable cause. Measurement of the blood's 'thickness' (ability to clot) in the operating theatre helps identify the cause and can both indicate the best treatment and monitor the body's response to that treatment.

This study will evaluate the ability of a new measurement device using high frequency sound (ultrasound) rebounding from a tiny sample of clotting blood to demonstrate different types of clotting disorder, and to compare it's accuracy to an existing device that works by measuring the stickiness of blood as it clots in a small cup. It will also compare the ability of both devices to match the surgeon's visual assessment of bleeding and clot formation in the surgical wound.

A recent National Institute of Clinical Excellence guideline (DG13 - 2014) acknowledges that standard laboratory screening tests are of limited diagnostic value in the setting of cardiac surgery owing both to delays in obtaining results and to their frequent inability to distinguish between causes of abnormal clotting. This guidance recommends point-of-care tests that measure changes mechanical strength of blood clot over time ("viscoelastic testing"), such as the TEG6 device. The new Quantra device measures similar changes in the physical properties of clotting blood using ultrasound, and has recently shown promising results in cardiac surgery. In this setting it appears to help distinguish between low levels of the clotting factor fibrinogen and low platelets as causes of impaired clotting, and may be superior to the TEG6. The present study will assess clotting in a group of patients with more severe clotting abnormalities and much heavier bleeding, and the benefits seen in cardiac surgery may be more marked.

Patients having major abdominal organ transplants (liver and liver-intestine transplants) typically have heavy bleeding, as much as all the blood in the body (about 5 litres) many times over (up to 30 litres or more). This is replaced continuously with donated or recycled blood and clotting factors to keep the patient alive, but frequent blood testing is essential. This is to identify what treatments are needed to maintain normal function of the heart, lungs, kidneys and other organs, and normal blood clotting. Blood samples are taken from special tubes or 'lines' routinely placed in blood vessels while the patient is asleep before surgery begins. When bleeding occurs during surgery special clotting factors and drugs can be given to improve clotting and help reduce bleeding, but these can have harmful effects, so the types and doses need to be guided by the results of clotting tests.

Routine blood sampling during these procedures consists of 15 ml (3 tsp) taken every 60 minutes 5-10 times during the operation. In this study, an extra 6 ml (1.2 tsp) will be taken at the same times and from the same lines as these standard samples, allowing us to study the clotting measurements in the new Quantra device and compare these to similar measurements in another theatre-based device already in routine use, as well as to standard clotting tests done in the laboratory. At times of sampling the operating surgeon will also give a score indicating the state of blood clotting from visual assessment of the internal surfaces exposed by the surgery. The two devices' measurements of clotting, laboratory tests and the visual score given by the surgeon will be compared to assess the best indicator of the severity of the bleeding and response to treatment.

The patient will not be managed differently from normal routine in any way apart from the small additional amounts of blood (maximum of 15-60 ml, or 3 -12 tsp) needed for Quantra measurements. No treatments will be based on these measurements.

ELIGIBILITY:
Inclusion Criteria: Sequential adult liver and multi visceral transplant recipients -

Exclusion Criteria: None envisaged

-

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult liver and multi visceral transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Quantra® parameters' correlation with conventional laboratory tests (including thrombin generation), TEG® 6S parameters and clinical bleeding scores. | 1 year
  Quantra® parameters:
  CT (clot time, intrinsic pathway) CS (clot stiffness) FCS (fibrinogen contribution to clot stiffness) PCS (platelet contribution to clot stiffness) Fibrinolysis Index
  TEG® 6S parameters:
  TEG-ACT (activated clotting time) R-time (reaction time) K-time (coagulation time) Alpha angle (clot formation) Maximum Amplitude (clot strength) LY30 (clot lysis % at 30 minutes) FLEV / Functional Fibrinogen (fibrinogen concentration)
  +/- Endogenous Thrombin Potential (thrombin generation)
  Surgeon's visual rating of clinical coagulopathy (Trans-Agency Consortium for Trauma Induced Coagulopathy (TACTIC) scoring system, adapted for liver transplantation): 0 (exceptionally dry surgical field) to 5 (very oozy with no visible clot); +/- perceived 'surgical' element: none, partial, mostly surgical), to be performed at times of routine sampling.

CONTACTS AND LOCATIONS:
Overall Officials: John R Klinck, FRCPC, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data can be shared with other investigators on request, at PI's and sponsor's discretion.